CLINICAL TRIAL: NCT01895257
Title: A Randomised Phase III Trial Comparing Hepatic Arterial Injection of Yttrium-90 Resin Microspheres (SIR-spheres) Plus Systemic Maintenance Therapy Versus Systemic Maintenance Therapy Alone for Patients With Unresectable Liver Metastases From Colorectal Cancer Which Are Controlled After Induction Systemic Therapy
Brief Title: Comparing HAI-90Y (SIR-spheres)+Chemotx LV5FU2 Versus Chemotx LV5FU2 Alone to Treat Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Prof. Marc Peeters, Professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The SIR-step trial; 2012-000508-14 (EudraCT Number)
Record Dates: First submitted 2013-06-06; First posted 2013-07-10 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Cancer
Keywords: TTP1; TTP2; PFS; Safety; R0 resection rate; Quality of life; Overall Survival
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Levoleucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: systemic chemotherapy LV5FU2 alone (Active Comparator): Modified LV5FU2 as described in protocol (6.2.1) D1-2 +/- bevacizumab or cetuximab or panitumumab (according its previous use) every 2 weeks
  Interventions: Drug: systemic chemotherapy LV5FU2
- B:SIR-spheres+systemic chemotherapy LV5FU2 (Active Comparator): ARM B: (Hepatic Arterial Infusion) HAI-90Y radioembolization (SIR-spheres injection) + modified LV5FU2 +/- bevacizumab or cetuximab or panitumumab according its previous use (refer to protocol).
  Interventions: Device: HAI-90Y radioembolization (SIR-spheres injection)

INTERVENTIONS:
Device: HAI-90Y radioembolization (SIR-spheres injection) — Patients randomised to receive the combination of SIR-Spheres microspheres plus systemic chemotherapy LV5FU2 need to be assessed in order to determine their suitability for SIRT.
  1. Hepatic Angiogram
  2. Liver-Lung Break-Through Nuclear Scan
  Other Names: Sir-spheres microspheres; SIRT
  Arms: B:SIR-spheres+systemic chemotherapy LV5FU2
Drug: systemic chemotherapy LV5FU2 — Systemic chemotherapy with modified LV5FU2 will be administered according to the following regimen.
  Cycle 1 onwards:
  Day 1 Hour 0: Leucovorin L (levoleucovorin) 200 mg/m2 (or folinic acid 400 mg/m²) in 250 ml glucose 5%, 2-hour IV infusion Hour + 2: 5-FU bolus 400 mg/m2, IV bolus Hour + 2: 5-FU continuous infusion 2400 mg/m2, 46-hour cont. IV infusion Day 14 End of cycle. To be repeated every 14 days until evidence of treatment failure.
  Other Names: Leucovorin L; Levoleucovorin; 5-FU; 5-Fluoro-Uracil
  Arms: A: systemic chemotherapy LV5FU2 alone

SUMMARY:
The investigators propose to conduct a randomised phase III trial evaluating a maintenance strategy comparing hepatic arterial injection of Yttrium-90 resin microspheres plus continuing simplified chemotherapy with/without targeted therapy versus continuing simplified chemotherapy with/without targeted therapy alone for patient with dominant or exclusive and unresectable liver mCRC controlled after 3-6 months of chemotherapy induction.

DETAILED DESCRIPTION:
The aim of the study is to investigate whether an intensified maintenance treatment of SIRT + simplified maintenance chemotherapy has a benefit in terms of time to progression (TTP) compared to simplified chemotherapy maintenance alone, in patients with stable disease after 3-6 months induction therapy. We would like to demonstrate the feasibility and safety of this approach and to investigate if this strategy has the potential to increase the outcome of the patient.

Primary end-point:

- Time to first progression (TTP1 overall)

Secondary end-points:

* Time to global progression (TTP1 + TTP2), Time to second progression (TTP2), TTP1 liver only
* Progression Free Survival (PFS)
* Overall Survival (OS)
* Safety
* Ro resection rate
* Quality of Life

Exploratory analysis:

- Prediction and evaluation of SIR-spheres treatment response (only for Belgian centres)

ELIGIBILITY:
Inclusion criteria:

1. Willing and able to provide written informed consent
2. Histologically confirmed adenocarcinoma of the colon or rectum, with or without primary tumour in situ. Unequivocal and measurable (RECIST 1.1) CT evidence of liver metastases which are not treatable by surgical resection and/or local ablation with curative intent at the time of trial entry.
3. Partial response or stable disease (RECIST 1.1 criteria, controlled metastatic disease) after chemotherapy induction with oxaliplatin and/or irinotecan based induction chemotherapy (doublet or triplet combinations) +/- targeted therapies during 3 to 6 months.
4. Trial inclusion must be performed between 3 and 6 months since the date of the first course of chemotherapy (induction) administration.
5. Limited extra-hepatic metastases in the lung and/or lymph nodes are permitted. Metastases in the lung must either be not more than five nodules in number with no individual nodule more than 1 cm in diameter or 1 single lesion of up to 1.7 cm in diameter. Involvement of lymph nodes in 1 single anatomic region (pelvis, abdomen or chest) are permitted provided their longest diameter measures less than 2 cm.
6. All imaging evidence used as part of the screening process must be within 28 days prior to the time of randomisation.
7. Suitable for either treatment regimen as determined by clinical assessment undertaken by the Investigator.
8. Patients may have received adjuvant chemotherapy or (neo-) adjuvant chemo-radiotherapy to the pelvis, provided the last dose of chemotherapy was administered at least 6 months prior to begin chemotherapy induction. Previous radiotherapy to the pelvis is not an exclusion criterion.
9. WHO performance status 0 - 1
10. Adequate hematological, renal and hepatic function as follows:

    Hematological Neutrophils > 1.5 x 109/L Platelets > 100 x 109/L Renal Creatinine < 1.5 x ULN (Upper Limit Normal) Hepatic Bilirubin ≤ 1.0 X ULN Albumin ≥ 30g/L ALT ≤ 5.0 x ULN AST ≤ 5.0 x ULN LDH ≤ 2.5 x ULN The date of blood tests must be within 28 days prior to the time of randomisation.
11. Age 18 years or older.
12. Female patients must either be postmenopausal, sterile (surgically or radiation- or chemically-induced), or if sexually active using an acceptable method of contraception.
13. Male patients must be surgically sterile or if sexually active and having a pre-menopausal partner must be using an acceptable method of contraception.
14. Life expectancy of at least 3 months without any active treatment.

Exclusion criteria

1. Evidence of ascites, cirrhosis, portal hypertension, main portal venous tumour involvement or thrombosis as determined by clinical or radiological assessment.
2. More than 6 months since last chemotherapy administration before trial inclusion.
3. Previous radiotherapy delivered to the upper abdomen.
4. Non-malignant disease that would render the patient unsuitable for treatment according to this protocol.
5. Prior major liver resection: remnant liver < 50% of the initial liver volume. Patient with a biliary stent can be included.
6. Liver tumor involvement > 80% before study inclusion (not at diagnosis but when trial inclusion for the patient is planned).
7. Resectable metastatic disease at trial inclusion.
8. Progressive disease during first-line metastatic chemotherapy. Adjuvant chemotherapy for colorectal cancer is not an exclusion criterion provided that it was completed more than 6 months prior to start of 1st line chemotherapy.
9. No oxaliplatin or irinotecan use during the first 3 to 6 months induction chemotherapy.
10. Pregnant or breast feeding.
11. Concurrent or prior history of cancer other than adequately treated non melanoma skin cancer or carcinoma in situ of the cervix.
12. Severe allergy to non-ionic contrast agents which would prevent contrast media use during the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP1 overall) | Up to 36 months
  Time to first progression (TTP1 overall)

SECONDARY OUTCOMES:
Time to global progression (TTP1 + TTP2) | Up to 42 months
  - Time to global progression (TTP1 + TTP2), Time to second progression (TTP2), TTP1 liver only
PFS | Up to 42 months
  Progression free survival
Safety | Up to 42 months
R0 resection rate | Up to 42 months
Quality of life | Up to 42 months
  Using
  * EORTC QLQ C30
  * EQ-5D
Overall Survival (OS) | Up to 42 months

OTHER OUTCOMES:
SIR-spheres treatment | Up to 42 months
  Prediction and evaluation of SIRspheres treatment response (only for Belgian sites)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Peeters, Study Chair — Universiteit Antwerpen; Marc Van den Eynde, Study Chair — University of St-Luc
Locations (10):
- Belgium (10):
  - University of Antwerp, Edegem, Antwerp
  - ASZ Aalst, Aalst
  - Institut Jules Bordet, Brussels
  - CUB Hôpital Erasme, Brussels
  - University of St-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - ZOL Genk, Genk
  - AZ St-Lucas Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHU de Liège, Liège